CLINICAL TRIAL: NCT07019961
Title: Comparison of the GMA-TULIP and I-gel Laryngeal Mask for Airway Management in General Anaesthesia: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KYLL-202502-002-01
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03

CONDITIONS: Trauma Surgery; General Anesthesia
Keywords: GMA-TULIP laryngeal mask; i-gel laryngeal mask; anatomical alignment of laryngeal mask; oropharyngeal leak pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G group (Experimental): Participants who will use the GMA-TULIP laryngeal mask
  Interventions: Device: the GMA-TULIP laryngeal mask
- I Group (Active Comparator): Participants who will use the i-gel laryngeal mask
  Interventions: Device: the i-gel laryngeal mask

INTERVENTIONS:
Device: the GMA-TULIP laryngeal mask — insert GMA-TULIP laryngeal masks after anesthesia induction
  Arms: G group
Device: the i-gel laryngeal mask — insert i-gel laryngeal masks after anesthesia induction
  Arms: I Group

SUMMARY:
The goal of this clinical trial is to learn if GMA-TULIP laryngeal mask willfit well in the right place in participants undergoing trauma surgery in a supine position under general anaesthesia.

It will also learn about the convenience, effectiveness and safety of the GMA-TULIP laryngeal mask.

The main questions it aims to answer are:

Does the GMA-TULIP laryngeal mask exhibit better anatomical alignment? Does the GMA-TULIP laryngeal mask perform effectively in trauma surgery patients in a supine position under general anaesthesia? Researchers will compare with the i-gel laryngeal mask (a device already popular among anaesthetists) to see if the GMA-TULIP laryngeal mask works to have a good performance in general anaesthesia.

Participants will describe feelings immediately after anesthesia， 1 hour later and 24 hours later.

ELIGIBILITY:
Inclusion Criteria:

18 years old ≤ age ≤ 70 years old. Patients undergoing trauma surgery in a supine position under general anesthesia.

18 kg/m2 ≤ BMI ≤ 35 kg/m2. American Society of Anesthesiologists (ASA) grades I-III. Can understand the research process and the use of pain scales. Clear understanding and voluntary participation in the study, signing of informed consent form.

Exclusion Criteria:

Patients with known or predicted difficult airways. High risk of reflux or aspiration (e.g., gastroesophageal reflux disease patients).

Individuals with active upper respiratory tract infections. Cervical related diseases or surgical history. Preoperative sore throat or previous sore throat or hoarseness. Patients with oral and maxillofacial trauma or fractures. Other reasons why researchers believe it is not appropriate to participate in the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of anatomical alignment under fiberoptic bronchoscopy observation | After insertion of laryngeal mask
  Class I: Vocal cords visible. Class II: Vocal cords and posterior epiglottis visible. Class III: Vocal cords and anterior epiglottis visible, <50% visual obstruction of epiglottis to vocal cords.
  Class IV: Vocal cords and anterior epiglottis visible, >50% visual obstruction of epiglottis to vocal cords.
  Class V: Vocal cords not visible. We define Class I and II field of view as accurate alignment; Class III and IV vision are defined as poor alignment; Class V vision is defined as alignment failure.

SECONDARY OUTCOMES:
Number of laryngeal mask insertions | After anesthesia induction
Placement time of laryngeal mask | After anesthesia induction
Difficulty level of laryngeal mask insertion | After insertion of laryngeal mask
Time of insertion of gastric tube through laryngeal mask airway | After insertion of laryngeal mask
Number of gastric tube insertions | After insertion of laryngeal mask
Difficulty level of gastric tube insertion | After insertion of laryngeal mask
Oral and pharyngeal leakage pressure | 10 minutes after stable ventilation and 1 hour after ventilation
Accuracy of anatomical alignment under fiberoptic bronchoscopy observation | 1 hour after ventilation and at the end of surgery
Success rate of initial ventilation placement | During the anesthesia process
Success rate of intraoperative ventilation | During the anesthesia process
Number of laryngeal mask adjustments during surgery | During the anesthesia process
Intraoperative injury situation | During the surgical process
Postoperative respiratory complications | Immediately after anesthesia awakening, 1 hour later, 24 hours later

CONTACTS AND LOCATIONS:
Overall Officials: Shaozhong Yang, Doctor, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
After the research is completed, share research data, research plans, statistical analysis plans, informed consent forms, and other data
Supporting Information: Study Protocol, SAP, ICF, CSR